CLINICAL TRIAL: NCT07147387
Title: Lions Hearts: A Community Approach to Multigenerational Cardiovascular Disease Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Janette Watkins, Assistant professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00027631
Record Dates: First submitted 2025-08-08; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular (CV) Risk

STUDY DESIGN:
Intervention Model Description: This study uses a two-arm, parallel-group design with a waitlist control. Mother-child dyads are allocated to either the immediate intervention group or a waitlist control group. The intervention group participates in a 12-week family-based physical activity program, delivered in community CrossFit affiliate settings. Sessions occur twice weekly and include functional strength and cardiovascular training, flexibility exercises, goal-setting, and family-oriented health education. The waitlist control group receives the same 12-week intervention following completion of all post-assessments. Both groups complete baseline, mid-intervention, post-intervention, and 3-month follow-up assessments to evaluate physical activity, health behaviors, cardiovascular fitness, and psychosocial outcomes. This design allows for evaluation of feasibility, acceptability, and preliminary effectiveness of the intervention while ensuring all participants have access to the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Control): Waitlist (Delayed Lion Hearts Program) (No Intervention): Participants in this group will serve as a waitlist control and will not receive the intervention during the initial study period. They will continue with their usual activities and will be offered the Lion Hearts program after the completion of the trial.
- Lion Hearts Physical Activity Program (Experimental): Participants in this group will take part in Lion Hearts, a community-based physical activity program delivered in partnership with local CrossFit affiliates. The program uses high-intensity functional training (HIFT) and family-based co-design strategies to promote cardiovascular health and increase moderate-to-vigorous physical activity among mothers and their children.
  Interventions: Behavioral: Lion Hearts Family-Based Physical Activity Program

INTERVENTIONS:
Behavioral: Lion Hearts Family-Based Physical Activity Program — The Lion Hearts Family-Based Physical Activity Program is a 12-week, community-based intervention designed to improve cardiovascular health and physical activity behaviors among mother-child dyads. The program consists of twice-weekly, 60-minute group exercise sessions delivered at local CrossFit affiliates. Each session includes scalable functional movement exercises, strength training, cardiovascular conditioning, and flexibility activities appropriate for both adults and children. In addition to physical activity, sessions incorporate goal-setting, family teamwork activities, and health education components to promote sustainable behavior change. The program was co-designed with community members during earlier study phases and is tailored to support engagement, feasibility, and family bonding.
  Arms: Lion Hearts Physical Activity Program

SUMMARY:
This pilot study evaluates the feasibility, acceptability, and preliminary effectiveness of Lion Hearts, a community-based, family-centered physical activity intervention designed to improve cardiovascular health among mother-child dyads. Developed through community co-design, the 12-week intervention is delivered in local CrossFit affiliates and includes twice-weekly fitness sessions incorporating functional movement, goal setting, teamwork, and health education. The study aims to assess changes in physical activity, fitness, and cardiovascular health markers, as well as family dynamics and motivation for physical activity. Participants complete baseline, mid-, post-, and 3-month follow-up assessments, including surveys, fitness testing, accelerometry, and optional lab work. Findings will inform the refinement of the intervention for future large-scale trials.

DETAILED DESCRIPTION:
The Lion Hearts study is a three-phase, community-based research project designed to reduce multigenerational cardiovascular disease (CVD) risk through a family-centered physical activity intervention. This record describes Phase 3, a pilot trial evaluating the feasibility, acceptability, and preliminary effectiveness of the Lion Hearts intervention among mother-child dyads.

The intervention was co-designed during Phase 2 using implementation mapping with mothers, children, certified fitness professionals, and community stakeholders. In Phase 3, the refined intervention will be delivered over 12 weeks in community fitness settings, specifically local CrossFit affiliates. The program consists of twice-weekly, 60-minute family fitness sessions, which include functional strength and cardiovascular exercises scaled appropriately for adults and children. Sessions also integrate components of goal setting, teamwork, and health education to foster family bonding and promote sustainable behavior change.

Participants will complete comprehensive assessments at four time points: baseline (Weeks 1-2), mid-intervention (Week 6), post-intervention (Weeks 13-14), and 3-month follow-up. Assessments include:

Surveys measuring physical activity, health behaviors, quality of life, and family functioning Fitness assessments (e.g., cardiovascular endurance, strength, flexibility) Physical health markers (e.g., height, weight, waist circumference, blood pressure) 7-day physical activity monitoring using accelerometers Optional laboratory bloodwork (e.g., lipid profiles, glucose levels) Semi-structured interviews and focus groups to evaluate participant experience and program acceptability The pilot trial will assess key implementation outcomes (feasibility, fidelity, satisfaction, and attendance), as well as preliminary signals of effectiveness on physical activity behavior, cardiovascular health, and psychosocial outcomes. The findings will guide further adaptation and inform the design of a larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Mother-child dyad willing to participate together in the full 12-week intervention and assessment activities
* Child aged 10-17 years old
* Mother (or female caregiver)
* Both mother and child must be able to safely engage in moderate-to-vigorous physical activity, as determined by pre-participation health screening (e.g., PAR-Q+)
* Access to transportation to attend twice-weekly exercise sessions at a local CrossFit affiliate

Exclusion Criteria:

* Presence of a medical condition that would make participation in moderate-to-vigorous physical activity unsafe, as determined by health screening or medical provider (e.g., uncontrolled hypertension, cardiovascular disease, severe orthopedic limitations)

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Mother (or female caregiver) Any gender child
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity - FitBit | Baseline (within 1 week prior to intervention start) and immediately post-intervention (within 1 week after completing the 12-week program).
  Physical activity behavior will be assessed using Fitbit wearable activity monitors for 7 days pre-intervention and 7 days post-intervention. Fitbits use accelerometry and heart rate sensors to estimate daily time spent in different intensity categories. The primary outcome will be minutes of moderate-to-vigorous physical activity (MVPA) per day, derived from Fitbit activity intensity classifications. Secondary measures include total step counts and sedentary time.
Retention rate of program | Immediately post-intervention (within 1 week after completing the 12-week program).
  percentage of eligible participants enrolled
Implementation fidelity of program | Immediately post-intervention (within 1 week after completing the 12-week program).
  percentage of planned sessions delivered, based on facilitator checklists
Participant adherence to program | Immediately post-intervention (within 1 week after completing the 12-week program).
  percentage of study requirements completed, based on attendance logs and completion of assessments
Recruitment rate of program | Immediately post-intervention (within 1 week after completing the 12-week program).
  percentage of eligible participants enrolled
Bioelectrical Impedance Analysis (BIA) | Baseline (within 1 week prior to intervention start) and immediately post-intervention (within 1 week after completing the 12-week program).
  Bioelectrical Impedance Analysis (BIA) is a non-invasive method used to estimate body composition, including fat mass, lean body mass, and total body water. The technique works by sending a safe, low-level electrical current through the body and measuring the resistance (impedance) encountered by the current. Because lean tissue contains more water and conducts electricity better than fat tissue, impedance values can be used to calculate body composition using validated prediction equations.

SECONDARY OUTCOMES:
submaximal cycle ergometer test - cardiovascular fitness | Baseline (within 1 week prior to intervention start) and immediately post-intervention (within 1 week after completing the 12-week program).
  Aerobic capacity will be assessed using a submaximal cycle ergometer test. Participants complete a graded exercise protocol on a stationary bicycle, during which workload and heart rate responses are recorded. Using validated prediction equations, these data are used to estimate maximal oxygen uptake (VO₂ max), a gold-standard indicator of cardiorespiratory fitness.
Exercise Regulations Questionnaire - BREQ-3 | Baseline (within 1 week prior to intervention start) and immediately post-intervention (within 1 week after completing the 12-week program).
  The Exercise Regulations Questionnaire (BREQ-3) is a validated self-report instrument designed to assess behavioral regulations for exercise based on Self-Determination Theory. The BREQ-3 measures the degree to which individuals are motivated to engage in physical activity across a continuum from amotivation to intrinsic motivation. The 24-item questionnaire includes six subscales: amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic regulation. Each item is scored on a 5-point Likert scale ranging from 0 ("Not true for me") to 4 ("Very true for me"). Subscale scores are calculated as the mean of relevant items, and higher scores indicate stronger endorsement of that form of regulation.
Barriers to Being Active Quiz | Baseline (within 1 week prior to intervention start) and immediately post-intervention (within 1 week after completing the 12-week program).
  The Barriers to Being Active Quiz is a standardized instrument developed by the Centers for Disease Control and Prevention (CDC) to identify perceived barriers that may prevent individuals from engaging in regular physical activity. The 21-item questionnaire assesses seven categories of barriers: lack of time, social influence, lack of energy, lack of willpower, fear of injury, lack of skill, and lack of resources. Each category is represented by three items, and responses are scored on a 4-point Likert scale ranging from 0 ("Very unlikely") to 3 ("Very likely").
Anxiety and Depression: Patient Health Questionnaire-4 | Baseline (within 1 week prior to intervention start) and immediately post-intervention (within 1 week after completing the 12-week program).
  The Patient Health Questionnaire-4 (PHQ-4) is an ultra-brief screening tool designed to assess core symptoms of anxiety and depression. It combines the two-item Generalized Anxiety Disorder scale (GAD-2) and the two-item Patient Health Questionnaire depression scale (PHQ-2) into a four-item measure. Each item is rated on a 4-point Likert scale from 0 ("Not at all") to 3 ("Nearly every day"), with total scores ranging from 0 to 12.
Social Support and Exercise Survey | Baseline (within 1 week prior to intervention start) and immediately post-intervention (within 1 week after completing the 12-week program).
  The Social Support and Exercise Survey is a validated instrument developed to measure the degree of support individuals perceive from family and friends for engaging in physical activity. The survey includes items that assess two domains of support: participation/encouragement (e.g., exercising together, offering reminders) and rewards/punishments (e.g., criticism or discouragement). Respondents indicate how often specific supportive or unsupportive behaviors occurred during the past three months using a 5-point Likert scale ranging from 1 ("None") to 5 ("Very often").
Body Appreciation Scale-2 (BAS-2) | Baseline (within 1 week prior to intervention start) and immediately post-intervention (within 1 week after completing the 12-week program).
  The Body Appreciation Scale-2 (BAS-2) is a validated self-report measure designed to assess positive body image. The 10-item questionnaire captures individuals' acceptance, respect, and appreciation of their bodies, as well as their ability to resist unrealistic appearance ideals promoted in society. Items are rated on a 5-point Likert scale ranging from 1 ("Never") to 5 ("Always"), with total scores calculated as the mean of all items.
Multidimensional Assessment of Interoceptive Awareness | Baseline (within 1 week prior to intervention start) and immediately post-intervention (within 1 week after completing the 12-week program).
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a validated self-report questionnaire designed to measure multiple dimensions of interoceptive body awareness. The MAIA assesses how individuals perceive, interpret, and respond to bodily sensations across eight subscales: Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening, and Trusting. Items are rated on a 6-point Likert scale from 0 ("Never") to 5 ("Always"), with higher scores indicating stronger interoceptive awareness in each domain.
Basic Psychological Needs Satisfaction and Frustration Scale | Baseline (within 1 week prior to intervention start) and immediately post-intervention (within 1 week after completing the 12-week program).
  The Basic Psychological Needs Satisfaction and Frustration Scale (BPNSFS) is a validated self-report instrument grounded in Self-Determination Theory. It assesses the extent to which individuals experience satisfaction and frustration of the three universal psychological needs: autonomy (feeling a sense of choice and control), competence (feeling effective and capable), and relatedness (feeling connected to others). The scale includes parallel subscales for both satisfaction and frustration, with items rated on a 5-point Likert scale ranging from 1 ("Not true at all") to 5 ("Completely true").

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
This is a small-scale pilot feasibility trial, and the dataset is not sufficiently powered or generalizable for meaningful secondary analyses. In addition, the dataset contains sensitive family- and health-related information, which poses a risk of re-identification even with standard de-identification procedures.